CLINICAL TRIAL: NCT03706053
Title: Midodrine Use for Hypotension Requiring IV Vasopressor Therapy in Early Septic Shock
Brief Title: Midodrine Use in Septic Shock
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding for the study; not enough staff
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Alexandra Kadl, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20889
Record Dates: First submitted 2018-09-26; First posted 2018-10-15 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized to intervention or placebo by the investigational pharmacy. Care providers, investigators and participants will be blinded to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Investigational pharmacy formulated placebo. In early phase patients will be randomized to placebo, 10mg TID midodrine or 20 mg TID midodrine. (15 per group)
  Interventions: Other: placebo
- Midodrine Hydrochloride 10 mg TID (Experimental): In early phase patients will be randomized to placebo, 10mg TID midodrine or 20 mg TID midodrine. (15 per group). After the first 45 patients are enrolled, interim safety and efficacy analysis will dictate which experimental group is continued/open to further enrollment (either 10 mg midodrine TID or 20 mg midodrine TID).
  Interventions: Drug: Midodrine Hydrochloride
- Midodrine Hydrochloride 20 mg TID (Experimental): In early phase patients will be randomized to placebo, 10mg TID midodrine or 20 mg TID midodrine. (15 per group). After the first 45 patients are enrolled, interim safety and efficacy analysis will dictate which experimental group is continued/open to further enrollment (either 10 mg midodrine TID or 20 mg midodrine TID).
  Interventions: Drug: Midodrine Hydrochloride

INTERVENTIONS:
Drug: Midodrine Hydrochloride — Midodrine Hydrochloride, enteral, 10 or 20 mg
  Arms: Midodrine Hydrochloride 10 mg TID; Midodrine Hydrochloride 20 mg TID
Other: placebo — investigational pharmacy formulated placebo comparator
  Arms: Placebo

SUMMARY:
The investigators aim to perform a randomized, double-blind, placebo-controlled trial to investigate the efficacy of midodrine in decreasing time to IV vasopressor liberation in patients with septic shock.

DETAILED DESCRIPTION:
A growing body of literature comprising largely retrospective data seems to support the safety and efficacy of midodrine in the intensive care unit for decreasing IV vasopressor use. The investigators hypothesize that administration of midodrine in the early phase of septic shock in patients with adequate enteral access will result in a significant decrease in time to IV vasopressor liberation (increase in vasopressor-free days), secondarily resulting in decreased central venous catheter dwell times and intensive care unit length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18-89 years old
* Admitted to UVA medical ICU with diagnosis of septic shock.
* Patients requiring at least 5 mcg/min norepinephrine infusion (or equivalent) for blood pressure support for at least 3 hours
* Patients with enteral access established within 12 hours of admission (either able to swallow, or feeding tube in place)

Exclusion Criteria:

* Pregnant females; (due to the potential adverse effects to an unborn child); patients with childbearing potential will have results of pregnancy test checked (which is routinely performed on admission); should the patient have child-bearing potential and the pregnancy status is not checked as part of routine care, such patients will be excluded from the study (i.e. pregnancy testing will not be performed for research purposes)
* Patients < 18 years
* Prisoners
* Patients already taking midodrine
* Patients with cirrhosis of the liver as defined by either biopsy, imaging findings of cirrhosis AND thrombocytopenia or patients otherwise undergoing liver transplant evaluation
* Patients with Increased intraocular pressure and glaucoma
* Patients with allergy to midodrine
* Non-English speaking patients, due to the narrow time-frame for study enrollment and execution of study protocol, employing interpreters is deemed to be a significant burden on the investigators with potential to hamper study enrollment. Non-english speaking patients are not deemed to be adversely affected by exclusion from study as there is no clear a priori reason why study results would not also apply to non-English speakers.
* Patients without enteral access within 12 hours of initiation of IV vasopressors
* Patients where the attending physician does not clinically intend to target a mean arterial pressure of > 65 mmHg
* Patients with pheochromocytoma or thyrotoxicosis
* Patients with active bowel ischemia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kadl, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Started | 3 | 4 | 3
Completed | 3 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID | Total
Number analyzed (Participants) | 3 | 4 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 2 | 2 | 1 | 5
Age, Continuous [Mean (Full Range); unit: years] | 65 [55 to 72] | 65.5 [57 to 75] | 62.33 [53 to 73] | 65.4 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 2 | 3 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 2 | 3 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Days Free of Vasopressors (Days)
Description: days without vasopressor adjusted with mortality
Time Frame: 90 days from enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
days | 24.3 [24 to 25] | 7.5 [0 to 27] | 25.6 [24 to 27]

2. Secondary Outcome: Central Venous Catheter Free Days
Time Frame: 90 days from enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
days | 15.3 [0 to 23] | 7.25 [0 to 28] | 25 [23 to 28]

3. Secondary Outcome: Intensive Care Unit Length of Stay (ICU LOS; Days)
Time Frame: 90 days from enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
days | 6 [5 to 7] | 10 [1 to 23] | 7.6 [5 to 10]

4. Secondary Outcome: Hospital Length of Stay (Hospital LOS; Days)
Time Frame: 90 days from enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
days | 11.3 [8 to 17] | 11 [1 to 23] | 15.7 [10 to 26]

5. Secondary Outcome: 30-day Mortality
Time Frame: 30 days from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
Participants | 2 | 1 | 0

6. Secondary Outcome: 90-day Mortality
Time Frame: 90 days from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
Participants | 2 | 1 | 0

7. Secondary Outcome: In-hospital Mortality
Description: Mortality during sentinel admission
Time Frame: From randomization until date of death if occurred prior to discharge from sentinel hospitalization, assessed up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
Participants | 1 | 1 | 0

8. Secondary Outcome: Intensive Care Unit Mortality
Description: Mortality during intensive care unit stay during sentinel admission
Time Frame: From randomization until date of death if occurred prior to discharge from the sentinel intensive care unit admission, assessed up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
Participants | 1 | 1 | 0

9. Secondary Outcome: Need to Re-initiate IV Vasopressors 2 or More Hours After Discontinuation
Time Frame: From randomization until date of discharge from the sentinel intensive care unit admission, assessed up to 52 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
Number analyzed (Participants) | 3 | 4 | 3
participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 30 days. All-Cause Mortality was assessed from randomization until date of discharge from the sentinel intensive care unit admission, up to 52 weeks.
Description: Adverse event data were collected for 30 days. All-Cause Mortality was assessed from randomization until date of discharge from the sentinel intensive care unit admission, with follow-up for up to 52 weeks. Two subjects died in the ICU. One additional subject died within 30 days of ICU admission but had been discharged prior.
Arm/Group | Placebo | Midodrine Hydrochloride 10 mg TID | Midodrine Hydrochloride 20 mg TID
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03706053/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT03706053/ICF_001.pdf